CLINICAL TRIAL: NCT00814242
Title: A Randomized Control Trial of Hepatectomy Versus Radiofrequency Ablation for Hepatocellular Carcinoma Adjacent to Major Blood Vessels
Brief Title: Hepatectomy Versus Radiofrequency Ablation for Hepatocellular Carcinoma Adjacent to Major Blood Vessels
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospotal, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHBH-RCT-2008-009
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Adjacent to Major Blood Vessels; Surgical resection; Ppercutaneous radiationfrequency ablation; Time to recurrence; Disease-free survival; Overall survival
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hepatectomy (Active Comparator): Patients with HCC adjacent to major blood vessels recieved radical resection.
  Interventions: Procedure: surgical resection
- percutaneous radiationfrequency ablation (Experimental): CT or Ultrasound-guided percutaneous radiofrequency ablation
  Interventions: Procedure: percutaneous radiationfrequency ablation

INTERVENTIONS:
Procedure: surgical resection — radical resection performed in patinets with HCC.
  Other Names: hepatectomy group
  Arms: hepatectomy
Procedure: percutaneous radiationfrequency ablation — CT or Ultrasound-guided percutaneous radiofrequency ablation performed in patinets with HCC
  Other Names: PRFA Goup
  Arms: percutaneous radiationfrequency ablation

SUMMARY:
This study will compare and analyze the difference between hepatectomy at deep and complex sites(adjacent to major blood vessels) of patients with HCC and PRFA prognosis, recovery after treatment as well as incidence of complications so as to establish treatment standards of HCC at these sites.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC), a serious disease with high incidence at home and abroad still shows a rising trend. In recent decade, the overall survival rate of the disease has entered a platform stage with little advance despite diversified methods of treatment. The prognosis of HCC is not so satisfying. In recent years, lots of clinical practice and a small amount of evidence-based medicine show that: ①.Surgical treatment is still the preferred choice of the treatment of HCC. ②. The standardization of comprehensive treatment should be put in top priority in current treatment of HCC. Rational treatment methods should be adopted in accordance with specific conditions of patients. The best and latest treatment methods should also be provided to improve the efficacy to the largest extent for the benefit of the majority of patients with HCC.

Today, tumor remaining in a patient after therapy with curative intent(eg. surgical resection for cure ) is categorized by a system known as R classification. That is shown: RX: presence of residual tumor can not be assessed; R0: no residual tumor; R1: microscopic residual tumor; R2: macroscopic residual tumor; The residue with the application of R classification not only refers to both residual tumor at the margin of surgical excision but also residue in distant metastasis. The higher R classification is, the worse the prognosis becomes.

Most studies have been leaded a good result By now that percutaneous radiationfrequency ablation(PRFA) is efficacious and safe for patients with HCC. In patients with HCC smaller than 3cm, PRFA may be comparable to suegical resection in long-term outcome.

At present, radical resection (for the final R0 or R1) performed in HCC at most deep and complex sites (including caudate lobe HCC, 8th segment hepatoma adjacent to the trunk of inferior vena cava, hepatic vein and portal vein, etc) often lead to serious damage to major blood vessels (i.e., hepatic vein, short hepatic vein, portal vein and inferior vena cava) and hemorrhage during surgery. Therefore, when the surgeon performs surgery near major sites, he should excise as few normal liver tissues as possible to avoid above-mentioned hazard. However, the resection margin may not be complete and thus affect radical effect. In addition, as the tumor is rather deep located, lots of normal liver tissues on the surface of the tumor are excised with massive bleeding and serious damage. In view of this situation, the surgeon will adopt some alternatives (PRFA is rather common) to achieve the efficacy similar to liver excision and greatly reduce the risk of vascular injury and some complications like hepatic insufficiency. However, there are no studies on the efficacy comparison between this treatment method and the efficacy of liver excision, time to recurrence (TTR)stage, disease-free survival and overall survival condition.

This study will compare and analyze the difference between hepatectomy at deep and complex sites of patients with HCC and PRFA prognosis, recovery after treatment as well as incidence of complications so as to establish treatment standards of HCC at these sites.

ELIGIBILITY:
Inclusion Criteria:

* Identify patients with HCC in accordance with the clinical diagnostic criteria of HCC passed at the Chines Eighth National Live Cancer Academic Conference. Patients with HCC shall be diagnosed with pathology. There is at least one measurable lesion.
* Hepatoma involved in this research at complex site is located at the eighth segment of liver, the substantial depth of liver below hepatic integument adjacent to the trunk of inferior vena cava, hepatic vein and portal vein. The tumor is located at hepatic caudate lobe. The maximal diameter < or=3m, AJCC/UICC-TNM stage is stage II and above. Lesions are determined by three senior hepatobiliary experts independently, therefore radical resection is possible. There is no possibility of extra-hepatic metastasis and tumor thrombus of portal vein, hepatic vein, vena cava and bile duct.
* Criteria of liver function: Child A level, serum bilirubin ≤ 1.5 times the upper limit of normal value, alanine aminotransferase and aspartate aminotransferase ≤ 2 times the upper limit of normal value. It's appropriate to perform liver resection and minimally invasive treatment.
* No dysfunction in major organs; Blood routine, kidney function, cardiac function and lung function are basically normal.
* Patients who can understand this trial, male or female, aged 18-70 voluntarily participate in clinical trials and have signed information consent.

Exclusion Criteria:

* Patients with apparent cardiac, pulmonary, cerebric and renal dysfunction,which may affect the treatment of liver cancer.
* Patients with other diseases which may affect the treatment mentioned here.
* Patients with medical history of other malignant tumors.
* Subjects participating in other clinical trials.
* Women in pregnancy and breast-feeding.
* Patients with tumor AJCC/UICC-TNM stage at IIIA period or below.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
tumor recurrence rate in one or two years; Disease-free survival;Overall survival. | 1,2,or 3 years

SECONDARY OUTCOMES:
Overall survival rate in one, two，three or five years; Disease-free survival in one, two，three or five years; hepatic function of patients after surgery, the incidence rate of complications and the decline level of serum AFP concentration. | one, two，three or five years

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shen, M.D., Study Chair — Eastern Hepatobiliary Surgery Hospital, Second Military Medical University
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality, China